CLINICAL TRIAL: NCT04863001
Title: Adescriptive Study on the Use of Antiarrhythmic Drugs in Pediatrics Cardiology Unit Assiut University
Brief Title: Use of Antiarrhythmic Drugs in Pediatrics
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Areej Tarek Mostafa mohamed makhlouf, Principle investegator , Areej Tarek Mostafa, Assiut University
Other Study IDs: antiarrhythmic drugs in pediat
Record Dates: First submitted 2021-04-14; First posted 2021-04-28 (Actual); Last update posted 2021-05-06 (Actual); Status verified 2021-04

CONDITIONS: Antiarrhythmic Toxicity
MeSH Terms: interventions — Anti-Arrhythmia Agents

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Antiarrhythmic drug — all classes of antiarrhythmic drugs used in pediatrics cardiology unit assiut university

SUMMARY:
This study aims to describe the use of Cardiovascular Drugs in Pediatrics Cardiology unit Assiut University. As regard :

* indications of use .
* proper dosage.
* proper management of side effects of their use.

DETAILED DESCRIPTION:
Arrhythmias occur in children and adolescents with congenital heart disease as well as those with structurally normal hearts. Antiarrhythmic medications primarily affect the ion channels in cardiac myocytes that are responsible for generating currents that create the action potential.

By altering the activity of these ion channels, the action potential is changed in an attempt to reduce the likelihood of sustained arrhythmias. There is awide range of antiarrhysmic drugs used in treatment Antiarrhysmics are therefore divided into five classes

Class I: Antiarrhythmics that affect sodium channels (slow depolarization) Class II: Drugs that counteract the sympathetic nervous system, predominantly beta-blockers Class III: drugs that affect the potasium channels ( prolong repolarization) Class IV: Drugs that affect calcium channels (Calcium channel blockers) Class V: Vagotonic drugs (Digoxin) and other miscellaneous drugs

ELIGIBILITY:
Inclusion Criteria:

* All Patients with Arrhythmic cardiac diseases admitted at cardiology unit Assiut University Hospital aged from 1 month to 18 years

Exclusion Criteria:

* ● Patients with diseases rather than arrhythmic cardiac diseases

Ages: 1 Month to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: 1- Patients' selection:- patients from 1 month age till 18 years on antiarrhythmic medications in Cardiology Unit Assiut University Hospital antiarrhytmic medications .
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
descripe the use of antiarrhythmic drugs in pediatrics | one year
  to asses the use of antiarrhythmic drugs in cardiology unit whether its used for proper indications matching with last guidelines or not to asses also dosage (gram per Kg of weight) of each drug used .and detrimine the side effects appear and its proper management.
  * proper dosage.
  * proper management of side effects of their use

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Podrid PJ. Antiarrhythmic drug selection. Annu Rev Med. 1987;38:1-17. doi: 10.1146/annurev.me.38.020187.000245. PMID 3555284